CLINICAL TRIAL: NCT00809185
Title: A Phase 2 Trial of RAD001(Everolimus) in Low and Intermediate-1 Risk Myelodysplastic Syndrome
Brief Title: RAD001(Everolimus) in Treating Patients With Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1905; P30CA043703 (NIH); CASE-CCF-8514 (Other: Cleveland Clinic IRB); CASE1905 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2012-05-04 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-02

CONDITIONS: Myelodysplastic Syndromes
Keywords: de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; previously treated myelodysplastic syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Everolimus; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 (everolimus) (Experimental): RAD001 (everolimus) at 10mg/day with Bone marrow aspirate/biopsy and other laboratory biomarker analysis
  Interventions: Drug: everolimus; Other: laboratory biomarker analysis; Procedure: Bone marrow aspirate/biopsy

INTERVENTIONS:
Drug: everolimus — Patients will receive monotherapy with RAD001(everolimus)for 21 days within the 28 day cycle.
  Other Names: RAD001
Other: laboratory biomarker analysis — Laboratory correlates (cytotoxic t cell populations, S6K1 levels, GSTT-1 mutations, and the presence or absence of HLA-DR15) will be assessed to see if any of these correlates correspond to response.
Procedure: Bone marrow aspirate/biopsy — Bone marrow aspirate and biopsy with cytogenetics should be obtained within 4 weeks prior to starting drug and at week 33. A bone marrow aspirate and biopsy should also be obtained for patients going off study prior to week 33 (including cytogenetics). The percentage of blasts on the aspirate should be used to determine the IPSS score.

SUMMARY:
RATIONALE: RAD001(Everolimus) may stop the growth of cancer cells by blocking some of the enzymes needed for their growth and by blocking blood flow to the cancer.

PURPOSE: This phase II trial is studying how well RAD001(everolimus) works in treating patients with myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical activity (improvement in erythroid response and/or improvement in other cytopenias, bone marrow morphology/cytogenetics) of RAD001(everolimus) in patients with low or intermediate-1 risk myelodysplastic syndromes.
* Assess the toxicity of this drug in these patients.

Secondary

* Examine laboratory correlates (S6K1 levels, angiogenesis pre- and post-treatment) and determine how these correlates correspond to dosing and clinical activity of RAD001(everolimus).
* Evaluate the presence of HLA-DR15 and cytotoxic T-cell populations in patients pre- and post-treatment and correlate this with response to treatment.
* Examine the incidence of the null GSTT-1 phenotype in myelodysplastic syndromes patients and correlate this with response to RAD001(everolimus).

OUTLINE: Patients receive oral RAD001(everolimus) once daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or relapse.

Blood samples are collected periodically during study. Samples are analyzed for S6K1 activity, effector T cells by flow cytometry, GSTT-1 by PCR, and HLA-DR15 levels.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Low or intermediate-1 risk myelodysplastic syndromes by International Prognostic Scoring System (IPSS) criteria

  * IPSS score < 1.5
* Requiring transfusion of 2 units of red blood cells at least once a month (four weeks prior to accrual on study)
* High levels of endogenous epoetin alfa (i.e., > 200 mU/mL)

  * Unlikely to respond to epoetin alfa, or has a documented clinical non-response to epoetin alfa (at a dose of ≥ 40,000 U weekly) or darbepoetin alfa (at a dose > 200 mcg every other week) (i.e., < 2 g/dL increase in hemoglobin and no decrease in transfusion requirements after at least 4 weeks of treatment)
* No chronic myelomonocytic leukemia

PATIENT CHARACTERISTICS:

* ECOG Performance Status of 0-2
* Liver enzymes (AST and ALT) and total bilirubin ≤ 2 times upper limit of normal
* Serum creatinine ≤ 2 times upper limits of normal
* No clinically significant anemia due to iron, B12, or folate deficiencies; autoimmune or hereditary hemolysis; or gastrointestinal bleeding
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious or poorly controlled medical condition that could be exacerbated by or complicate compliance with study therapy

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior treatment (including growth factors)
* No chronic use (> 2 weeks) of physiologic doses of a corticosteroid agent (dose equivalent to > 10 mg/day of prednisone) within 28 days of the first day of study drug
* No concurrent use of another investigational agent
* No concurrent therapy with any cytotoxic drugs, steroids, or growth factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-11; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Advani, MD, Study Chair — Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Advani AS, Mahfouz RZ, Maciejewski J, Rybicki L, Sekeres M, Tripp B, Kalaycio M, Bates J, Saunthararajah Y. Ribosomal S6 kinase and AKT phosphorylation as pharmacodynamic biomarkers in patients with myelodysplastic syndrome treated with RAD001. Clin Lymphoma Myeloma Leuk. 2014 Apr;14(2):172-177.e1. doi: 10.1016/j.clml.2013.10.001. Epub 2013 Nov 11. PMID 24332215

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Cleveland Clinic medical hospital from April 2006-March 2009
Groups:
- RAD001(Everolimus): drug will be administered at 10mg by mouth for 21 days followed by a 7 day rest period
Period: Overall Study
Arm/Group | RAD001(Everolimus)
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RAD001(Everolimus)
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 67 [60 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Either a Major or Minor Erythroid Response (Hemoglobin Change From Baseline Measure)
Description: Major erythroid response: (1) For patients with a baseline hemoglobin less than 11 g/dL, a major erythroid response is defined as a > 2 g/dL increase in hemoglobin from baseline; or (2) 100% decrease in red blood cell transfusion requirements.
  Minor erythroid response: (1) For patients with baseline hemoglobin less than 11 g/dL, a minor erythroid response is defined as an increase in hemoglobin greater than 1 g/dL but less than 2 g/dL from baseline; or (2) > 50% decrease in red blood cell transfusion requirements.
Time Frame: 2 years of treatment
Population: All patients enrolled and given treatment.
Measure: Number; unit: participants
Arm/Group | RAD001(Everolimus)
Number analyzed (Participants) | 7
participants
  Number of Patients with a Minor Response | 0
  Number of Patients with a Major Response | 0

2. Secondary Outcome: Number of Dose- and Non-dose-limiting Toxicities
Description: Number of Dose- and Non-dose-limiting Toxicities at the end of cycle 1 associated with RAD001 (see AE/SAE section for details).
Time Frame: at end of one cycle (28 days)
Population: All patients enrolled and given treatment.
Measure: Number; unit: events
Arm/Group | RAD001 (Everolimus)
Number analyzed (Participants) | 7
events | 26

3. Secondary Outcome: Number of Participants With Bone Marrow Morphology and Cytogenetics Pre- and Post-therapy
Description: Number of Participants with change in bone marrow morphology and cytogenetics
Time Frame: at 2 years of treatment
Population: All patients enrolled and given treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | RAD001(Everolimus)
Number analyzed (Participants) | 7
Participants | 0

4. Other Pre Specified Outcome: Laboratory Correlates (Cytotoxic T-cell Populations, S6K1 Levels, GSTT-1 Mutations, and Presence or Absence of HLA-DR15)
Description: T-cell populations in patients pre- and post-treatment
Time Frame: at 2 years of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were measure during treatment which ranges from 5-196 days.
Arm/Group | RAD001(Everolimus)
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001(Everolimus) (N=7)
infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001(Everolimus) (N=7)
bleeding (General disorders) | 2
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
fatigue (General disorders) | 3
fever/infection (Infections and infestations) | 4
neutropenia (Blood and lymphatic system disorders) | 3
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
rash (Skin and subcutaneous tissue disorders) | 1
renal insufficiency (Renal and urinary disorders) | 1
stomatitis (Infections and infestations) | 2
thrombocytopenia (Blood and lymphatic system disorders) | 3
weight loss (General disorders) | 2

LIMITATIONS AND CAVEATS:
The trial was stopped early due to slow accrual. 18-33 patients were needed to address objectives, however only 7 patients were enrolled. Insufficient patients responded to the treatment to allow laboratory correlates with response to be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes